CLINICAL TRIAL: NCT00649610
Title: Randomized, Double Blind, Multicenter Study of the Safety and Efficacy of Valdecoxib 40 mg Once Daily vs. Diclofenac 75 mg Twice Daily in Subjects With Acute Low Back Pain
Brief Title: Randomized, Double Blind, Multicenter Study of the Safety and Efficacy of Valdecoxib 40 mg Once Daily Compared With Diclofenac 75 mg Twice Daily in Acute Low Back Pain
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: A3471012
Record Dates: First submitted 2008-03-28; First posted 2008-04-01 (Estimated); Last update posted 2008-04-10 (Estimated); Status verified 2008-03

CONDITIONS: Low Back Pain
Keywords: acute low back pain
MeSH Terms: conditions — Low Back Pain | interventions — valdecoxib; Diclofenac

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 (Active Comparator)
  Interventions: Drug: valdecoxib
- Arm 2 (Active Comparator)
  Interventions: Drug: diclofenac

INTERVENTIONS:
Drug: valdecoxib — valdecoxib 40 mg QD for 7 days with a second dose of 40 mg the first day
  Arms: Arm 1
Drug: diclofenac — diclofenac 75 mg twice daily (BID) for 7 days
  Arms: Arm 2

SUMMARY:
The pain relief, safety, and tolerability of valdecoxib 40 mg once daily compared with diclofenac 75 mg twice daily for acute low back pain was studied. The effect of valdecoxib on the patient's level of disability and quality of life was also studied.

ELIGIBILITY:
Inclusion Criteria:

* Acute low back pain, defined as either class 1a or class 2a according to the Quebec Task Force Classification and categorized as moderate-severe in the Pain Intensity Categorical Scale and Visual analogue score (VAS) greater or equal to 50 mm
* Acute low back pain was to have started at least 72 hours prior to inclusion in the trial and more than 6 weeks after the last episode of acute low back pain
* History of at least 1 reported episode of acute low back pain in the last 5 years

Exclusion Criteria:

* History of inflammatory arthritis, chronic pain, metastasis, Paget's disease, or other diseases known to cause pain
* Moderate to severe scoliosis
* Back pain due to major trauma or visceral disorder
* Unwilling to refrain from commencing concomitant physiotherapy
* Active or suspected esophageal, gastric pyloric channel, or duodenal ulceration or bleeding within 30 days prior to the first dose of study medication
* Any known laboratory abnormality, which in the opinion of the investigator, would contraindicate study participation
* Subject was pregnant or lactating woman , or was a woman of childbearing potential not using an acceptable method of contraception

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 340 (Actual)
Dates: Start 2002-11; Study Completion 2003-05 (Actual)

PRIMARY OUTCOMES:
Subject-rated VAS Pain Intensity (0 - 100 mm), which was evaluated using the change from baseline | Day 3

SECONDARY OUTCOMES:
Patient global evaluation | Day 3 and Day 7
Subject's functional capacity as measured by the Oswestry Low Back Pain and Disability Questionnaire | Day 7
Subject's quality of life as measured by the Acute short form (SF)-36 (8 domains) | Day 7
Pain Relief | Day 3 and Day 7
Composite Upper Gastrointestinal (UGI) Tolerability was calcluated. A subject had a UGI event if the subject reported at least 1 of the following: moderate or severe nausea, or moderate or severe abdominal pain, or moderate or severe dyspepsia | Day 7
VAS Pain Intensity (0-100 mm) | Day 7
Categorical Pain Intensity | Day 3 and Day 7

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (19):
- Argentina (2):
  - Pfizer Investigational Site, Bs. As.
  - Pfizer Investigational Site, Buenos Aires
- Brazil (4):
  - Pfizer Investigational Site, Goiânia, Goiás
  - Pfizer Investigational Site, Curitiba, Paraná
  - Pfizer Investigational Site, Petrópolis, Rio de Janeiro
  - Pfizer Investigational Site, São Paulo, São Paulo
- Pfizer Investigational Site, Santiago, Chile
- Colombia (3):
  - Pfizer Investigational Site, Bogotá, D.C.
  - Pfizer Investigational Site, Bogota D.C
  - Pfizer Investigational Site, Cali-valle
- Costa Rica (2):
  - Pfizer Investigational Site, Cartago, Cartago Province
  - Pfizer Investigational Site, Hatillo Centro, Provincia de San José
- Pfizer Investigational Site, Quito, Pichincha, Ecuador
- Mexico (3):
  - Pfizer Investigational Site, Toluca, EDO. de Mexico
  - Pfizer Investigational Site, Zapopan, Jalisco
  - Pfizer Investigational Site, Puebla City, Puebla
- Pfizer Investigational Site, Lima, Lima Province, Peru
- Venezuela (2):
  - Pfizer Investigational Site, Caracas, DF
  - Pfizer Investigational Site, Caracas

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A3471012&StudyName=Randomized%2C%20Double%20Blind%2C%20Multicenter%20Study%20of%20the%20Safety%20and%20Efficacy%20of%20Valdecoxib%2040%20mg%20Once%20Daily%20Compared%20With%20Diclofenac%2075%20